CLINICAL TRIAL: NCT00312247
Title: Biomechanical Analysis of Gait in Individuals With Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Michael D. Sussman, MD, Principal Investigator, Shriners Hospitals for Children
Other Study IDs: SHC-DMD-79115; SHC-79115 (Other Grant/Funding Number: Shriners Hospitals for Children)
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Walking; Muscle Strength; Energy Cost; Quality of Life
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Boys taking steroids: Boys who are taking prednisone or deflazacort
- Boys who are steroid naive: Boys who are not taking steroids for a variety of reasons

SUMMARY:
The purpose of this research study is to understand the walking patterns, strength and function changes of boys with Duchenne muscular dystrophy on/off corticosteroids to determine the best timing and treatment options to maintain walking for as long as possible.

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is an X-linked recessive disease of muscle characterized by a progressive loss of functional muscle mass, which is replaced with fibrofatty tissue. Historically, boys with DMD lose the ability to walk between the ages of 8-12 years, due to progressive weakness of the quadriceps coupled with the development of contractures at the hip, knee and ankle. This progressive loss in function necessitates individuals with DMD to spend less time walking and more time in wheelchairs, leading to the development of spinal deformities. Recently, corticosteroids have been shown to reduce the expected loss of muscle strength, extend the time that ambulation and standing are maintained, and minimize or eliminate spinal deformity in individuals with DMD; yet, the side effects of such treatment preclude use in some patients. To date, differences in gait patterns and other markers of disease progression between boys on corticosteroids and those not utilizing such treatment have not been objectively quantified. This lack of knowledge is a major obstacle to determining the most effective treatment for subsets of boys with DMD.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of DMD
* Male.
* Four years of age or older.
* Ability to walk independently for five minutes to 10 minutes at self-selected speed.
* Ability to cognitively understand directions for testing procedures.

Exclusion Criteria:

* Female
* Nonambulatory

Ages: 4 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Boys with DMD who are ambulatory starting at the age of 4 until ambulation ceases
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2006-04; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Gait pattern | every six months (2x/year)
  computerized assessment of walking

SECONDARY OUTCOMES:
muscle strength | every six months (2x/year)
  quantitative assessment of strength with a Biodex
energy cost of walking | every six months (2x/year)
  assessment of how much energy it takes to walk, assessed with a Cosmed K4b2
gross motor functional skills | every six months (2x/year)
  assessment of gross motor skills, ie getting up off the floor, ascending/descending stairs
Step activity Monitor-participation | one week every six months
  measurement of the number of steps taken in the community/home environment during weekdays and weekends

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Sussman, MD, Principal Investigator — Shriners Hospitals for Children
Locations (3):
- United States (3):
  - UCLA Department of Orthopaedic Surgery, Los Angeles, California
  - Shriners Hospitals for Children, Sacramento, California
  - Shriners Hospitals for Children, Portland, Oregon

REFERENCES:
- [Result] Sienko Thomas S, Buckon CE, Nicorici A, Bagley A, McDonald CM, Sussman MD. Classification of the gait patterns of boys with Duchenne muscular dystrophy and their relationship to function. J Child Neurol. 2010 Sep;25(9):1103-9. doi: 10.1177/0883073810371002. Epub 2010 Jun 29. PMID 20587736
- [Result] McDonald CM, McDonald DA, Bagley A, Sienko Thomas S, Buckon CE, Henricson E, Nicorici A, Sussman MD. Relationship between clinical outcome measures and parent proxy reports of health-related quality of life in ambulatory children with Duchenne muscular dystrophy. J Child Neurol. 2010 Sep;25(9):1130-44. doi: 10.1177/0883073810371509. Epub 2010 Jun 17. PMID 20558672
- See also: Shriners Hospitals for Children — http://www.Shrinershq.org